CLINICAL TRIAL: NCT06621238
Title: Effect of Musıc Lıstened to Prımarıparous Women Who Have Delıvered by Cesarean Sectıon on Paın, Status Anxıety and Breastfeedıng Success
Brief Title: The Effect of Musıc on Labor Paın, Anxıety and Breastfeedıng Success
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sibel ÖZTÜRK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ataturk University SOZTURK0005
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-09

CONDITIONS: Labor Pain; Anxiety; Breast Feeding; Post Operative Pain
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Breast Feeding; Pain, Postoperative | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vsisual Analog scale (VAS) (Experimental): It will be used to measure pain in the intervention and control groups during the postpartum period.
  Interventions: Behavioral: Music
- State anxiety scale (Experimental): It will be used to evaluate the mother's current anxiety status in the postpartum period.
  Interventions: Behavioral: Music
- Breastfeedıng Success (Experimental): It will be used to evaluate the breastfeeding success of mothers in the experimental and control groups in the postpartum period.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Listen to Music

SUMMARY:
The aim of this study is to examine the effects of music played to primiparous women who had a cesarean section on pain, state anxiety and breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* Caesarean section
* Live birth

Exclusion Criteria:

* Risky pregnancy
* Twin pregnancy
* Newborn with cleft palate, cleft lip

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study evaluates pain, state anxiety, and mothers' breastfeeding success in the postpartum period.
Enrollment: 140 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Postpartum Pain | Within the first hour after birth
  The Visual Analog Scale will be used to assess the level of cesarean pain in the postpartum period in the intervention and control groups. A minimum score of 1 and a maximum score of 10 are obtained from the scale. As the score obtained from the scale increases, it indicates that the pain also increases. After the pre-test and intervention, a change in pain and a change in the Visual Analog Scale score are expected in the intervention group.
State Anxiety | Within the first hour after birth
  The state anxiety scale evaluates the degree of severity of the emotions or behaviors experienced by the individual in the situation he/she is in. The highest score that can be obtained is 80, and the lowest score is 20. As the score obtained from the scale increases, it shows that the state anxiety also increases.
Breastfeeding Success | Within the first hour after birth
  The scale evaluates the success of mothers in breastfeeding their babies. The minimum score that can be obtained from the scale is 0 and the maximum score is 10, and a high score from the evaluation and diagnosis scale means that breastfeeding success is high.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel ÖZTÜRK, PhD, Principal Investigator — sibel.ozturk@atauni.edu.tr; Ayşegül ŞAHİSN ÇELEBİ, PhD, Principal Investigator — ascelebi@beu.edu.tr
Locations (1):
- Mardin Education and Research Hospital, Mardin, Artuklu/Mardin, Turkey (Türkiye)